CLINICAL TRIAL: NCT06004245
Title: A Phase I, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Anti-Tumor Activity of VVD-133214 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors Harboring Microsatellite Instability (MSI) and/or Deficient Mismatch Repair (dMMR)
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Anti-Tumor Activity of VVD-133214 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vividion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VVD-133214-01; 2023-503170-20-01 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Deficient mismatch repair; dMMR; Microsatellite instability; MSI
MeSH Terms: conditions — Microsatellite Instability | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open label study. Participants will be assigned to dose cohorts in the order in which they are enrolled. However, if two or more cohorts in the same part of the study are open for enrollment at the same time, participants will be randomized into these cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VVD-133214 Dose Escalation (Experimental)
  Interventions: Drug: VVD-133214
- VVD-133214 Monotherapy Expansion (Experimental)
  Interventions: Drug: VVD-133214
- VVD-133214 + Pembrolizumab Expansion (Experimental)
  Interventions: Drug: VVD-133214; Drug: Pembrolizumab

INTERVENTIONS:
Drug: VVD-133214 — VVD-133214 will be administered orally and once daily (QD) in 3-week cycles.
Drug: Pembrolizumab — Pembrolizumab will be administered by intravenous (IV) infusion at a fixed dose of 200 mg on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®
  Arms: VVD-133214 + Pembrolizumab Expansion

SUMMARY:
This is a first-in-human, Phase I, open-label, multicenter, dose-escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of VVD-133214 monotherapy, and in combination with pembrolizumab, in participants with microsatellite instability (MSI) and/or deficient mismatch repair (dMMR) advanced solid tumors. VVD-133214 is an oral drug that acts on a protein called Werner (WRN), which may promote the growth of cancers that are MSI and/or dMMR. By acting on WRN, VVD-133214 may be able to block the growth of these types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Have a microsatellite instability (MSI) and/or deficient mismatch repair (dMMR), histologically or cytologically documented advanced (unresectable and/or metastatic) solid tumor; for the combination with pembrolizumab only: Histologically confirmed locally advanced, or metastatic colorectal adenocarcinoma (CRC) with no prior systemic treatment for metastatic disease and not amenable to surgery
* Have received and then progressed following, or are intolerant to, standard therapy in the advanced setting
* Presence of measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Life expectancy of at least (≥)12 weeks
* Availability of formaldehyde-fixed paraffin-embedded (FFPE) archival tumor tissue for submission to Sponsor/central laboratory for retrospective central testing; for participants without archival tissue, a biopsy from either primary or metastatic tumor lesion, deemed medically feasible, must be taken
* Adequate hematologic, end-organ, and cardiovascular function, as defined in the protocol

Exclusion Criteria:

* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known hypersensitivity or intolerance to ingredients from the study drug formulation including patients with rare genetic disorders such as galactosaemia, glucose-galactose intolerance or congenital lactase deficiency
* Known uncontrolled central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control) and/or carcinomatous meningitis
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial (including but not limited to tuberculosis and atypical mycobacterial disease), parasitic, or other infection (excluding fungal infections of nail beds), or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization within 2 weeks prior to the start of drug administration (related to the completion of the course of antibiotics, except if for tumor fever) or 6 months for any intracranial abscess
* Has a positive test at screening for hepatitis B virus, hepatitis C virus, or for human immodeficiency virus (HIV), per local diagnostic standard and in accordance with local laws and regulations
* Uncontrolled diabetes or symptomatic hyperglycemia (i.e., well controlled defined as a screening hemoglobin A1c <8% and no urinary ketoacidosis)
* Significant cardiovascular/cerebrovascular disease within 6 months prior to Day 1 of study drug administration
* Alcohol or drug dependence or abuse
* Patients with known Werner (WRN) syndrome
* Prior treatment with any WRN helicase inhibitor
* Treatment with moderate or strong CYP3A4 inducers within 14 days prior to initiation of study treatment
* Treatment with moderate or strong CYP3A4 or P-glycoprotein inhibitors within 14 days prior to initiation of study treatment
* Pregnancy, breastfeeding, or intention of becoming pregnant during the study

Additional Exclusion Criteria for the Combination with Pembrolizumab Only:

* Active or history of autoimmune disease or immune deficiency with some exceptions
* History of interstitial lung disease or pneumonitis
* Treatment with systemic immunosuppressive medication (such as corticosteroids) within 2 weeks prior to initiation of study treatment with some exceptions
* Treatment with organ transplant/graft tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, with Severity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) | From first dose of study drug(s) until 30 days after the final dose of VVD-133214 or 90 days after last dose of pembrolizumab
Incidence of Dose-Limiting Toxicities | Cycle 1 (1 cycle is 3 weeks)

SECONDARY OUTCOMES:
Maximum Plasma Concentration Observed (Cmax) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Time of Maximum Plasma Concentration Observed (Tmax) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Area Under the Plasma Concentration-Time Curve (AUC) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Apparent Oral Clearance (CL/F) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Volume of Distribution (V/F) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Terminal Half-Life (T1/2) of VVD-133214 | At prespecified timepoints in Cycles 1, 2, and 3, and every 2 cycles thereafter (1 cycle is 3 weeks) until last dose of study drug (up to approximately 15 months)
Objective Response Rate | From start of study treatment until end of follow-up (up to approximately 36 months)
Disease Control Rate | From start of study treatment until end of follow-up (up to approximately 36 months)
Duration of Response | From the time of first occurrence of a documented response until the time of documented disease progression or death from any cause, whichever occurs first (up to approximately 36 months)
Progression-Free Survival, as Assessed by the Investigator | From start of study treatment to the first occurrence of documented disease progression or death from any cause, whichever occurs first (up to approximately 36 months)
Overall Survival | From start of study treatment to the time of death from any cause (up to approximately 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Vividion Therapeutics
Locations (25):
- United States (7):
  - City of Hope Cancer Center, Duarte, California
  - City of Hope - Santa Clarita, Valencia, California
  - Norton Cancer Institute - MDC, Louisville, Kentucky
  - Duke University, Durham, North Carolina
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Alfred Hospital, Melbourne, Victoria, Australia
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
- Rigshospitalet, København Ø, Denmark
- France (2):
  - CLCC Leon Berard Lyon, Lyon
  - Gustave Roussy, Villejuif
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona, BARCELONA
  - Clinica Universidad de Navarra Madrid, Madrid, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
- United Kingdom (3):
  - Sarah Cannon Research Institute, London
  - The Christie, Manchester
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: No